CLINICAL TRIAL: NCT06768528
Title: Association Between Galectin-3 and Post-operative AtrIal Fibrillation After Coronary Artery Bypass Graft
Acronym: GNOSIS
Status: Recruiting | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SDC 5346/21/121
Record Dates: First submitted 2022-12-20; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-12

CONDITIONS: Post-operative Atrial Fibrillation; Cardiovascular Diseases; Post-pericardiotomy Syndrome
Keywords: Post-operative atrial fibrillation; Galectin-3
MeSH Terms: conditions — Cardiovascular Diseases; Postpericardiotomy Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood sample for Galectin-3 dosage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Galectin-3 dosage — Peripheral blood sample will be collected in the 24h before CABG

SUMMARY:
The goal of this observational study is to test the association between high levels of Galectin-3 and the occurrence of post-operative atrial fibrillation after isolated coronary artery bypass grafting (CABG). The main question[s] it aims to answer are:

* Is Galectin-3 an accurate biomarker to predict higher risk of developing post-operative atrial fibrillation?
* Are high levels of Galectin-3 associated to other post-operative complications and major adverse cardiovascular events? Participants will be enrolled during pre-operative evaluation and a peripheral blood sample collection will be performed in the 24h before CABG. Participants will then be followed for a period of 12 months (daily during hospitalization and 3 appointments after hospital discharge) to determine whether patients with higher levels of Galectin-3 will have worse outcomes.

DETAILED DESCRIPTION:
Prospective, observational, single-center cohort study including patients undergoing coronary artery bypass graft (CABG) surgery.

Patients will be enrolled during preoperative evaluation. A peripheral blood sample will be collected within 24 hours before surgery and patients will be followed during hospitalization and for 12 months after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing coronary artery bypass graft surgery

Exclusion Criteria:

* Inability to sign the free and informed consent form
* Renal dysfunction with estimated glomerular filtration rate less than 30ml / min / 1.73m² or dialysis therapy
* Moderate to severe left ventricular dysfunction (ejection fraction < 40%)
* Patients with previous atrial fibrillation
* Pregnancy
* Concomitant valve surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Single-center cohort study with patients admitted for coronary artery bypass graft (CABG) surgery.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Galectin-3 and post-operative atrial fibrillation | Up to 7 days after surgery
  Evaluate the association of higher levels of Galectin-3 (in ng/mL) and the occurrence of post-operative atrial fibrillation lasting at least 12 hours or requiring cardioversion

SECONDARY OUTCOMES:
Galectin-3 and other post-operative complications | 6 weeks
  Evaluate the association of higher levels of Galectin-3 (in ng/mL) and the occurrence of post-operative complications, such as infection, bleeding, post-pericardiotomy syndrome, reoperation, systemic embolism, type 5 myocardial infarction
Galectin-3 and major adverse cardiovascular events | 12 months
  Evaluate the association of higher levels of Galectin-3 (in ng/mL) and the occurrence major adverse cardiovascular events, such as stroke, acute coronary syndrome, revascularization procedures and cardiovascular death
Galectin-3 and left atrial remodeling | 12 months
  Evaluate the association of higher levels of Galectin-3 (in ng/mL) and left atrial enlargement (both linear and volumetric echocardiographic measurements) and development of supraventricular arrhythmias in holter monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Leticia Carvalho, Principal Investigator — Instituto do Coração - HCFMUSP; Eduardo Lima, Study Director — Instituto do Coração - HCFMUSP
Locations (1):
- Instituto do Coração - Hospital das Clínicas - Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No